CLINICAL TRIAL: NCT00262093
Title: Angiogenesis Markers in Primiparas Versus Multiparas: Relevance to Preeclampsia Incidence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Other Study IDs: PRIMIMULTI-HMO-CTIL
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2005-11

CONDITIONS: Pre-Eclampsia
Keywords: preeclampsia; sFlt1; PlGF; parity; angiogenesis
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The reason for having a higher incidence of preeclampsia in primiparas may involve angiogenesis imbalance in these patients.

DETAILED DESCRIPTION:
Primiparity is one of the main risk factors for having preeclampsia during pregnancy. Recently, sFlt-1, soluble FMS-like tyrosine kinase-1, has been shown to be a major molecule involved in the pathogenesis of preeclampsia. Higher sFlt-1 mRNA, higher serum levels of sFlt-1 as well as lower PlGF, placental growth factor, have been found in preeclamptic patients.

We intend to check the angiogenesis profile of primiparas as compared to multiparas.

ELIGIBILITY:
Inclusion Criteria:

* Every delivery

Exclusion Criteria:

* Preeclampsia or pregnancy induced hypertension

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Bdolah, MD, MSc, Principal Investigator — Hadassah-Hebrew University Medical School
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel